CLINICAL TRIAL: NCT01301248
Title: Phase II Safety and Toxicity Study of Cisplatin With or Without Cetuximab and Concomitant Radiotherapy for Locoregionally Advanced Squamous Cell Carcinomas of the Head and Neck (SCCHN)
Brief Title: Cisplatin Chemoradiation With or Without Cetuximab for Locoregionally Advanced Squamous Cell Carcinomas (SCC) of the Head and Neck
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theagenio Cancer Hospital (Other Government)
Responsible Party: Charalambos Andreadis MD, PhD, Theagenio Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EEEK2008RCT2
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-04

CONDITIONS: Head and Neck Neoplasms; AJCC Stage III/IV
Keywords: locally advanced,; unresectable,; head and neck squamous cell carcinoma,; stage III/IV
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Chemoradiotherapy; Cetuximab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy/Cisplatin(GroupA) (Active Comparator): Radiotherapy 65-70 Gy (1.8 Gy fractionation) Chemotherapy delivered weekly (cisplatin; 40mg/m2)
  Interventions: Other: Chemoradiation
- Radiotherapy/Cisplatin/Cetuximab(GroupB) (Experimental): Radiotherapy 65-70 Gy (1.8 Gy fractionation) Chemotherapy delivered weekly (cisplatin; 40mg/m2)concurrently with weekly cetuximab 250mg/m2 (following initial loading dose of 400mg/m2 a week before radiotherapy initiation)
  Interventions: Other: Chemoradiation plus Cetuximab

INTERVENTIONS:
Other: Chemoradiation plus Cetuximab — Radiotherapy 65-70 Gy (1.8 Gy fractionation) Chemotherapy delivered weekly (cisplatin; 40mg/m2)concurrently with weekly cetuximab 250mg/m2 (following initial loading dose of 400mg/m2 a week before radiotherapy initiation)
  Other Names: Platinol; Erbitux
  Arms: Radiotherapy/Cisplatin/Cetuximab(GroupB)
Other: Chemoradiation — Radiotherapy 65-70 Gy (1.8 Gy fractionation) Chemotherapy delivered weekly (cisplatin; 40mg/m2
  Other Names: Platinol
  Arms: Radiotherapy/Cisplatin(GroupA)

SUMMARY:
To examine the safety and toxicity of concurrent radiotherapy with cisplatin with the further addition of cetuximab experimental treatment

DETAILED DESCRIPTION:
Conventional radiotherapy (65-70 Gy, 1.8 Gy per day) concurrently with weekly cisplatin (40mg/m2) (group A, n=25) or with weekly cisplatin (40mg/m2) and weekly cetuximab 250mg/m2, after initial dose of 400mg/m2) (group B, n=25) is applied (in a 1:1 randomization ratio). Groups will be matched age, sex, PS, and disease site.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed HNSCC of oral cavity, larynx, oropharynx or
* hypopharynx; age of 18 years or more
* adequate liver (SGOT, SGPT, ALP ≤ 3x normal)
* kidneys (creatinine clearance ≥ 60ml/min
* heart (no arrythmias, no heart failure) and
* bone marrow (WBC ≥ 4,000/μL, granulocytes ≥ 1,500/μL, Hb ≥ 10g/dL, platelets ≥ 100,000/μL) function
* ECOG performance status 0 or 1 and
* stage III or IVa to b with measurable lesions
* written informed consent

Exclusion Criteria:

* prior radiotherapy
* chemotherapy
* concurrent active malignancies
* pregnancy
* breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Determine safety and toxicity of combination | Time from first administration of trial treatment to death or last date known to be alive, anticipated average time frame 24 months
  Toxicity is graded according to National Cancer Institute Common Toxicity Criteria for Adverse Events version 1 system.

SECONDARY OUTCOMES:
Overall survival time | Time from first administration of trial treatment to death or last date known to be alive, anticipated average time frame 24 months
  Time from first administration of trial treatment to death. Patients without event are censored at the last date known to be alive or at the clinical cut-off date, whatever is earlier.
Progression-free survival time | Time from first administration of trial treatment to disease progression, death or last tumor assessment, anticipated average time frame 12 months
  Duration from first administration of trial treatment until progression (radiological or clinical, if radiological progression is not available) or death due to any cause. Patients without event are censored on the date of last tumor assessment.
Response | Time from first administration of trial treatment to disease progression, death or last tumor assessment, anticipated average time frame 12 months
  Complete response (CR) is defined as the total disappearance of radiographic evidence of tumour. Partial response (PR) is defined as the ≥50% reduction in the product of the maximal bidimensional tumour diameters. Stable disease defined any change between +25% and -50% in tumour size, and progressive disease included any increase >25% from baseline or the appearance of any new lesion. We record tumour shrinkage and time to the development of disease progression according to the revised RECIST criteria, v.1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Charalambos Andreadis, MD, Principal Investigator — Theagenio Cancer Hospital
Locations (1):
- Theagenio Cancer Hospital, Thessaloniki, Greece